CLINICAL TRIAL: NCT05644262
Title: Life's End Benefits of cannaBidiol and tetrahYdrocannabinol (LiBBY)
Brief Title: Life's End Benefits of cannaBidiol and tetrahYdrocannabinol
Acronym: LiBBY
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Medical University of South Carolina (Other); Alzheimer's Clinical Trials Consortium (Other); Alzheimer's Therapeutic Research Institute (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Paul S. Aisen, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATRI-007; R01AG068324 (NIH); R01AG095004 (NIH)
Record Dates: First submitted 2022-11-16; First posted 2022-12-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Agitation; Dementia
Keywords: agitation; hospice care-eligible; dementia; agitation and dementia (HAD); alzheimer's disease; alzheimer's disease dementia; alzheimer's disease and related dementias
MeSH Terms: conditions — Psychomotor Agitation; Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- T2:C100 (Experimental)
  Interventions: Drug: T2:C100
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: T2:C100 — The active study intervention, T2:C100, is an oral combination of tetrahydrocannabinol (THC) and cannabidiol (CBD) in a digestible oil. T2:C100 is a full spectrum oral solution with five non-reactive ingredients: delta-9-tetrahydrocannabinol (THC), cannabidiol (CBD), a pharmaceutical grade medium chain triglyceride (MCT) oil, and two flavoring agents (lemon and peppermint).
  During the double-blind treatment period, participants will receive 1mL study drug (T2:C100) twice daily for Baseline - Day 7 (approximately 1 week), and then will increase to 2mL study drug twice for the remainder of the double-blind treatment period (Day 7 - Week 12 (approximately 11 weeks)).
  Participants who enter the Open Label Extension will receive 1mL study drug (T2:C100) twice daily for Week 12 - Week 13 (approximately 1 week), and will then increase to 2mL study drug twice daily for the remainder of the Open Label Extension (Week 13 - Week 26 (approximately 23 weeks)).
  Other Names: TRC/CBD oral combination
  Arms: T2:C100
Drug: Placebo — Matching placebo in a digestible oil. The placebo contains only three non-reactive ingredients: medium chain triglyceride (MCT) oil and two flavoring agents (lemon and peppermint).
  During the double-blind treatment period, participants will receive 1mL placebo twice daily for Baseline - Day 7 (approximately 1 week), and then will increase to 2mL placebo twice for the remainder of the double-blind treatment period (Day 7 - Week 12 (approximately 11 weeks)).
  Arms: Placebo

SUMMARY:
This is a multicenter randomized double-blind placebo-controlled Phase 2 study of an oral combination of tetrahydrocannabinol (THC) and cannabidiol (CBD) compared to placebo over 12 weeks. This study is designed to test the hypothesis that treatment with an oral combination of THC/CBD will reduce agitation hospice care-eligible patients with agitation and dementia as measured by the Cohen Mansfield Agitation Inventory (CMAI) when compared to placebo at 2 weeks.

This study will enroll approximately 120 participants of any gender at least 40 years of age who are hospice care-eligible with agitation and dementia (HAD). Participants will be randomized (50:50) to either active study drug (T2:C100) or placebo.

The double-blind period of this study is 12 weeks. A 12 week optional open-label extension will be offered to participants who complete the double-blind period.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent from participant or legally authorized representative.
2. Person of any sex/gender 40 years of age or older.
3. Ability to take or be administered liquid medication.
4. Meets DSM-V criteria for Major Neurocognitive Disorder.
5. Current clinically significant agitation as demonstrated by an NPI-agitation subscale of 4 or above at Screening.
6. Meets at least one of the following requirements:

   1. Currently enrolled in out-patient or in-patient hospice care.
   2. Stage 6d on the Functional Assessment Staging Test (FAST).
   3. Score of 12 or more according to the Advanced Dementia Prognostic Tool (ADEPT) as implemented by the Mitchell Index.
7. Willing to agree not to use cannabinoids in any form (e.g., topically applied, ingested, inhaled, or other form of administration), other than the trial medication, during the first 12 weeks of the study.
8. Has a third-party clinician (e.g., hospice, palliative care, PCP) who is responsible for medical management of the participant outside the study.
9. In the opinion of the investigator, resides in an environment suitable to conduct a clinical trial (i.e., study intervention can be administered and concomitant medication use can be accurately documented).
10. In the opinion of the site PI, has a study partner (may be paid or unpaid caregiver) able and willing to provide accurate information about the participant, oversee the administration of study drug, and participate in study visits and informant-based assessments (usually requires at least 5 hours of contact per week).

    NOTE: Other knowledgeable informants/informed caregivers may contribute to informant-based scales; however, the site should identify an informant who will be able to serve as the primary source of information.
11. As assessed by investigator, participant is likely to be able to comply with the protocol for a minimum of 2 weeks.

Exclusion Criteria:

1. Use of cannabinoids or other forms of marijuana in the 3 weeks prior to Baseline, as based on self-report.
2. Suspected or known allergic reactions, adverse reactions, or hypersensitivity to cannabinoids and/or components (e.g., (<specify oil to be used in final formulation, e.g.: coconut oil; sesame oil>) of the study drug (T2:C100 or placebo).
3. Treatment with another investigational drug or other investigational intervention within the previous 30 days or five half-lives of the investigational product, whichever is longer.
4. Any condition, which in the opinion of the site PI, Data and Coordinating Center, regulatory sponsor, or Project Lead/Protocol PI, makes the participant unsuitable for inclusion.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in agitation as measured by the Cohen-Mansfield Agitation Inventory (CMAI) at 2 weeks | Baseline, Day 7 and Day 14
  The Cohen-Mansfield Agitation Inventory (CMAI) assesses the average frequency of manifestations of agitated behaviors in elderly persons over a 1-week period. The CMAI is a questionnaire consisting of 29 agitated behaviors, each rated on a 7-point frequency scale. In addition to the frequency of each behavior, informants/caregivers will be asked to use a 5-point scale to rate the disruptiveness of each behavior. For this study, the CMAI will target behaviors observed by knowledgeable informants/informed caregivers. Expanded descriptions of the behaviors will be provided to the informant/caregiver to be used as a reference during the interview.

SECONDARY OUTCOMES:
Change from Baseline in agitation as measured by the Cohen-Mansfield Agitation Inventory (CMAI) at 12 weeks | Baseline, Day 7, Day 14, Week 4, Week 8 and Week 12
  The Cohen-Mansfield Agitation Inventory (CMAI) assesses the average frequency of manifestations of agitated behaviors in elderly persons over a 1-week period. The CMAI is a questionnaire consisting of 29 agitated behaviors, each rated on a 7-point frequency scale. In addition to the frequency of each behavior, informants/caregivers will be asked to use a 5-point scale to rate the disruptiveness of each behavior. For this study, the CMAI will target behaviors observed by knowledgeable informants/informed caregivers. Expanded descriptions of the behaviors will be provided to the informant/caregiver to be used as a reference during the interview.
Clinical Global Impression of Change in Behavior (CGIC-B) | Baseline, Day 7, Day 14, Week 4, Week 8 and Week 12
  The Clinical Global Impression of Change in Behavior (CGIC-B) is similar to the mADCS-CGIC in that both versions provide a systematic method for assessing clinically significant change in clinical trials as evaluated by an experienced clinician on the basis of a clinical interview and examination. It relies on both direct examination and/or observation of the participant as well as interviews with a knowledgeable informant/informed caregiver. The participant interviews that are a part of the mADCS-GGIC are not feasible in this study population and have been eliminated in the CGIC-B in favor of standard administration across all participants. Anchors present in the mADCS-CGIC that are not relevant in this study population have been removed and agitation-related anchors have been added to the CGIC-B. A skilled and experienced clinician who is blinded to treatment assignment rates the patient on a 7-point Likert scale, ranging from 1 (marked improvement) to 7 (marked worsening).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Aisen, MD, Study Director — Alzheimer's Therapeutic Research Institute; Jacobo Mintzer, MD, Principal Investigator — Ralph H. Johnson Veterans Affairs Medical Center (VAMC); Brigid Reynolds, NP, Principal Investigator — Georgetown University
Locations (10):
- United States (10):
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Melgar-Caro Medcenter and Community Research (MCMCR), Miami, Florida
  - University of South Florida, Tampa, Florida
  - University of Kentucky, Lexington, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Case Western Reserve University, Beachwood, Ohio
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Vanderbilt University Medical Center Center for Cognitive Medicine, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- See also: ATRI Studies Page — https://atri.usc.edu/studies/
- See also: LiBBY Study Website — https://libbystudy.org/